CLINICAL TRIAL: NCT05207800
Title: Predictive Value of Maternal Serum Pentraxin 3 (PTX 3) and Heparin-binding Protein (HBP) for Chorioamnionitis in Preterm Premature Rupture of Membranes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2021-07-207
Record Dates: First submitted 2022-01-10; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Preterm Premature Rupture of Membrane
Keywords: pentraxin 3; heparin-binding protein; chorioamnionitis; preterm premature rupture of membranes; term premature rupture of membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Chorioamnionitis; Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy pregnant woman: healthy pregnant woman
  Interventions: Other: The concentrations of PTX3 and HBP were monitored in maternal blood, placental tissue and amniotic fluid.
- pregnant women with TPROM: pregnant women with term premature rupture of membranes
  Interventions: Other: The concentrations of PTX3 and HBP were monitored in maternal blood, placental tissue and amniotic fluid.
- pregnant women with PPROM: pregnant women with preterm premature rupture of membranes
  Interventions: Other: The concentrations of PTX3 and HBP were monitored in maternal blood, placental tissue and amniotic fluid.

INTERVENTIONS:
Other: The concentrations of PTX3 and HBP were monitored in maternal blood, placental tissue and amniotic fluid. — The concentrations of PTX3 and HBP were monitored in maternal blood, placental tissue and amniotic fluid.

SUMMARY:
Objective: The aim of this study was to investigate the predictive value of maternal serum pentraxin 3 (PTX3) and heparin-binding protein (HBP) for chorioamnionitis in preterm premature rupture of membranes (PPROM).

Method: This observational prospective cohort study included a total of 180 pregnant women at 24-40 gestational weeks. There were 60 cases of term premature rupture of membranes (TPROM), 60 cases of preterm premature rupture of membranes（PPROM）and 60 cases of healthy women. The concentrations of PTX3 and HBP were measured in maternal blood and amniotic fluid using an enzyme-linked immunosorbent assay (ELISA). Western immunoblotting was used to analyze the expression of PTX3 and HBP in placental tissue. The localization and immunoreaction of PTX3 and HBP in placenta were determined via immunohistochemistry (IHC).

ELIGIBILITY:
Inclusion Criteria:

1. The pregnant woman is born at a gestational age of 24-40 weeks;
2. The pregnant woman has a single child;
3. Regular obstetric examination during pregnancy with complete obstetric examination data was diagnosed as premature rupture of membranes (PROM).

Exclusion Criteria:

1. Pregnancy complicated with medical and surgical diseases, such as thyroid dysfunction and chronic hypertension;
2. Insufficiency of vital organ function or complicated tumor;
3. Pregnant women with other pregnancy complications besides PROM, such as preeclampsia, etc.;
4. Neonates had major congenital malformations (congenital anal atresia, congenital biliary atresia, congenital heart disease and so on, whether prenatal suspicion or diagnosis postpartum)
5. Neonatal septicemia, hemolytic disease or other diseases affecting bilirubin metabolism.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-02-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
PTX3 and HBP concentrations in maternal blood | 24 weeks to 40 weeks gestation
  PTX3 and HBP concentrations in maternal blood

SECONDARY OUTCOMES:
PTX3 and HBP concentrations in placental tissue | 24 weeks to 40 weeks gestation
  PTX3 and HBP concentrations in placental tissue

OTHER OUTCOMES:
PTX3 and HBP concentrations in amniotic fluid | 24 weeks to 40 weeks gestation
  PTX3 and HBP concentrations in amniotic fluid